CLINICAL TRIAL: NCT06544499
Title: A Phase 3, Multicenter, Randomized, Double-Blinded, Placebo-Controlled, Parallel-Arm Study Followed by an Open-Label Arm to Evaluate the Efficacy and Safety of Efgartigimod IV in Adult Participants With Primary Immune Thrombocytopenia
Brief Title: A Study to Assess the Efficacy and Safety of Efgartigimod IV in Adult Participants With Primary Immune Thrombocytopenia
Acronym: advance NEXT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-2402; 2024-515451-38-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-31; First posted 2024-08-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efgartigimod IV (Experimental): Participants receiving efgartigimod IV during the double-blinded treatment period and the open-label treatment period(s)
  Interventions: Biological: Efgartigimod IV
- Placebo IV (Experimental): Participants receiving placebo IV during the double-blinded treatment period and receiving efgartigimod IV during the open-label treatment period(s)
  Interventions: Biological: Efgartigimod IV; Other: Placebo IV

INTERVENTIONS:
Biological: Efgartigimod IV — Intravenous infusion of efgartigimod
Other: Placebo IV — Intravenous infusion of placebo
  Arms: Placebo IV

SUMMARY:
The main purpose of this study is to look at the effect (efficacy) and safety of efgartigimod IV in participants with primary immune thrombocytopenia (ITP). After an up to 2 weeks screening period, eligible participants will be randomized in a 2:1 ratio to receive either efgartigimod IV or placebo IV, respectively during the double-blinded treatment period (DBTP). At the end of the treatment period (up to 24 weeks), all participants will receive efgartigimod IV during the first 52-week open-label treatment period (OLTP1). At the end of the first OLTP1, participants may begin a second 52-week OLTP2. After the OLTP2, the participants will enter a follow-up period (approximately 8 weeks) while off study drug. The participants will be in the study for up to 138 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 18 years of age and the local legal age of consent for clinical studies when signing the informed consent form (ICF).
* Has documented baseline mean platelet count of <30 x 10^9/L before randomization
* Has a documented duration of primary immune thrombocytopenia (ITP) of more than 12 months on the date of informed consent form (ICF) signature.
* Has documented prior ITP treatment with at least 1 of the following treatments: corticosteroids, intravenous immunoglobulin (IVIg), anti-D immunoglobulin, thrombopoietin receptor agonist (TPO-RAs), or rituximab.
* Has documented insufficient response to a prior ITP treatment (the specific criteria can be found in the protocol).
* Has documented prior response defined as 1 platelet count of ≥50 × 109/L to at least 1 of the following ITP treatments in the 3 years before the date of ICF signature: prednisone, dexamethasone, other or nonspecified corticosteroids, IVIg, or anti-D immunoglobulin

Exclusion Criteria:

* Other than the indication under study, known autoimmune disease or any medical condition that would interfere with an accurate assessment of clinical symptoms of ITP, confound the results of the study or put the participant at undue risk.
* Secondary ITP
* Nonimmune thrombocytopenia
* Autoimmune hemolytic anemia
* ITP-associated critical or severe bleeding The complete list of criteria can be found in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Extent of disease control, defined as the number of cumulative weeks during the 24-week Double-Blinded Treatment Period with platelet counts of at least 50 × 10^9/L | Up to 24 weeks

SECONDARY OUTCOMES:
Proportion of participants achieving platelet counts of at least 50 × 10^9/L for at least 4 of the 6 study visits between study weeks 19 and 24 of the DBTP | Up to 6 weeks
Proportion of participants achieving platelet counts of at least 50 × 10^9/L for at least 6 of the 8 study visits between study weeks 17 and 24 of the DBTP | Up to 8 weeks
Proportion of participants achieving a platelet counts of at least 50 × 10^9/L for at least 8 of the 12 study visits between weeks 13 and 24 of the DBTP | Up to 12 weeks
Proportion of participants achieving a platelet count of at least 50 × 10^9/L on at least 4 occasions at any time until study week 12 during the DBTP | Up to 12 weeks
Time to response, defined as the time to achieve 2 consecutive platelet counts of at least 50 × 10^9/L at any time during the DBTP | up to 24 weeks
Proportion of participants with an IWG response during the DBTP | Up to 24 weeks
  International Working Group (IWG)
Proportion of participants with initial response, defined as a platelet count of at least 30 × 10^9/L and a 2-fold increase from baseline in platelet count at study week 5 of the DBTP | Up to 20 weeks
Time to achieve a platelet count of at least 30 × 10^9/L and a 2-fold increase from baseline in platelet count during the DBTP | Up to 24 weeks
Number of cumulative weeks during the DBTP with platelet counts of at least 30 × 10^9/L and ≥20 × 10^9/L above baseline | Up to 24 weeks
Number of cumulative weeks during the DBTP with platelet counts of at least 30 × 10^9/L and at least 20 × 10^9/L above baseline in participants with baseline platelet counts of <15 × 10^9/L | Up to 24 weeks
Extent of disease control, defined as the percentage of weeks with platelet counts of at least 50 × 10^9/L | Up to 76 weeks
In participants receiving placebo IV in the DBTP, the extent of disease control, defined as the number of cumulative weeks with platelet counts of at least 50 × 10^9/L | Up to 76 weeks
Overall platelet count response, defined as the proportion of participants achieving a platelet count of at least 50 × 10^9/L on at least 4 occasions during the first 52 weeks of treatment with efgartigimod IV | Up to 52 weeks
Mean change from baseline in platelet count at each study visit | Up to 76 weeks
The percentage of weeks with platelet counts of at least 30 × 10^9/L and at least 20 × 10^9/L above baseline | Up to 76 weeks
In participants with baseline platelet counts <15 × 10^9/L, the percentage of weeks with platelet counts of at least 30 × 10^9/L and at least 20 × 10^9/L above baseline | Up to 76 weeks
Proportion of participants who achieve a sustained platelet count response, defined as achieving platelet counts of at least 50 × 10^9/L for at least 4 occasions during 6-week intervals | Up to 76 weeks
In participants receiving placebo IV in the DBTP, the proportion of participants achieving platelet counts of at least 50 × 10^9/L for at least 8 of the 12 study visits between weeks 13 and 24 of the OLTP1 | Up to 12 weeks
In participants receiving placebo IV in the DBTP, proportion of participants who achieve sustained platelet count response, defined as achieving platelet counts of at least 50 × 10^9/L for at least 6 of 8 visits between weeks 17 and 24 of the OLTP1 | Up to 8 weeks
In participants receiving placebo IV in the DBTP, the extent of disease control, defined as the number of cumulative weeks with platelet counts of at least 50 × 10^9/L during the first 24 weeks of treatment with efgartigimod IV | Up to 24 weeks
Occurrence rate of rescue ITP therapy | Up to 76 weeks
Proportion of participants with reduction in concurrent ITP therapy during the OLTP1 | Up to 52 weeks
Incidence and severity of bleeding, assessed by the ITP Bleeding Scale (IBLS) | Up to 76 weeks
Incidence of AEs (including AEs of clinical interest) and SAEs | Up to 136 weeks
  AE = adverse event; SAE = serious adverse event; An adverse event of clinical interest is a pre-specified medically significant event that has the potential to be causally associated with the study drug.
Incidence of ADA against efgartigimod in serum over time | Up to 136 weeks
  ADA = antidrug antibodies
Incidence of NAb against efgartigimod in serum over time | Up to 136 weeks
  NAb = Neutralizing antibodies
Efgartigimod Cmax over time | Up to 136 weeks
Percent change from baseline in total IgG levels in serum over time | Up to 136 weeks
  IgG = immunoglobulin G

CONTACTS AND LOCATIONS:
Locations (92):
- United States (17):
  - Mayo Clinic Hospital Scottsdale, Phoenix, Arizona
  - University of Southern California Norris Comprehensive Cancer Center, Los Angeles, California
  - Sharp Memorial Hospital, Oceanside, California
  - University of Colorado Hospital, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - The University of Chicago Medicine, Chicago, Illinois
  - The University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Tulane University, New Orleans, Louisiana
  - Henry Ford Health, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Regional Cancer Care Associates, LLC (RCCA), Little Silver, New Jersey
  - Clinical Research Alliance Inc., Westbury, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University Hospital East, Columbus, Ohio
  - INTEGRIS Cancer Institute of Oklahoma, Oklahoma City, Oklahoma
- Austria (3):
  - Allgemeines Krankenhaus der Stadt Linz, Linz
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Klinikum Kreuzschwestern Wels, Wels
- Bulgaria (6):
  - Acibadem City clinic Tokuda hospital, Sofia
  - UMHAT Aleksandrovska, Sofia
  - University Multi-Profile Hospital for Active Treatment (UMHAT) St. Ivan Rilski, Sofia
  - National Specialized Hospital for Active Treatment of Hematology Diseases, Sofia
  - UMHAT SofiaMed, Sofia
  - University Hospital Prof. Dr. Stoyan Kirkovich AD, Stara Zagora
- China (11):
  - Beijing YouYi Hospital-Beijing Friendship Hospital Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - The First Affiliated Hospital Of Bengbu Medical College, Bengbu
  - The Affiliated Hospital of Chengde Medical University, Chengde
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - The Affiliated Huaian No.1 People's Hospital of Nanjing Medical University, Huai'an
  - Huizhou Central People's Hospital, Huizhou
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology (HUST), Wuhan
  - Wuxi People's Hospital (Wuxi No.1 People's Hospital), Wuxi
  - Affiliated Hospital of Jiangsu University, Zhenjiang
- University Hospital Center Zagreb, Zagreb, Croatia
- Czechia (2):
  - Fakultni Nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Kralovske Vinohrady, Prague
- France (3):
  - CHU d'Amiens-Picardie - Hopital SUD, Amiens
  - Centre Hospitalier Universitaire (CHU) - Hopital Henri Mondor, Créteil
  - Centre Hospitalier Universitaire Dijon Bourgogne Medecine Interne et Immunologie Clinique, Dijon
- Germany (2):
  - University Hospital Carl Gustav Carus, Dresden
  - Universitaetsklinikum Essen (AoR), Essen
- Hungary (2):
  - Semmelweis University-Internal Medicine and Haematology, Budapest
  - Gyor-Moson-Sopron Varmegyei Petz Aladar Egyetemi Oktato Korhaz, Győr
- Ireland (2):
  - Mater Misericordiae University Hospital, Dublin
  - St James's Hospital - Cancer Clinical Trials Office, Dublin
- Italy (11):
  - Azienda ULSS 7 Pedemontana, Bassano del Grappa
  - Universita Degli Studi Di Firenze - Azienda Ospedaliero-Universitaria Careggi (AOUC), Florence
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - AO Maggiore Della Carita, Novara
  - U.O.C. Ematologia Ospedale Santa Maria delle Croci, Ravenna
  - Arcispedale Santa Maria Nuova (ASMN) Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS), Reggio Emilia
  - A.O.U. Citta della Salute e della Scienza di Torino, Torino
  - AO Ordine Mauriziano di Torino, Torino
  - Azienda Sanitaria Universitaria Integrata, Trieste
  - ASST Sette Laghi Ospedale di circolo e Fondazione Macchi, Varese
- Poland (7):
  - Szpital Uniwersytecki nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Pratia Onkologia Katowice, Katowice
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
  - NZOZ Neuromed M. i M. Nastaj Sp.P., Lublin
  - Uniwersytecki Szpital Kliniczny Nr 4 w Lublinie Centrum Innowacyjnych Terapii, Lublin
  - Szpital Specjalistyczny im. Jedrzeja Sniadeckiego w Nowym Saczu, Nowy Sącz
  - Wojewodzki Szpital Zespolony im. Ludwika Rydygiera w Toruniu, Torun
- Portugal (2):
  - Unidade Local de Saude de Braga, Braga
  - Unidade Local de Saude Gaia e Espinho, E.P.E., Vila Nova de Gaia
- Romania (4):
  - Spitalul Clinic Coltea, Clinica de Hematologie, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic Judetean de Urgenta Sibiu (SCJS) (Clinical County Hospital Sibiu), Sibiu
  - Spitalul Clinic Judetean de Urgenta Targu-Mures, Târgu Mureş
- Serbia (5):
  - Clinical Center of Serbia, Belgrade
  - University Clinical Centre of Kragujevac, Kragujevac
  - Clinical Center of Nis, Niš
  - University Clinical Hospital Center Zemun, Zemun
  - General Hospital Djordje Joanovic, Zrenjanin
- Spain (6):
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - University Hospital Quironsalud Madrid, Pozuelo de Alarcón
  - Hospital Clinico Universitario - University of Valencia, Valencia
- United Kingdom (8):
  - Queen Elizabeth Hospital Birmingham - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Bradford Royal Infirmary - Bradford Teaching Hospitals NHS Foundation, Bradford
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Glasgow Royal Infirmary - North Glasgow University Hospital Division, Glasgow
  - University Hospitals of Leicester NHS Trust-Leicester Royal Infirmary, Leicester
  - Barts and the London Pathology & Pharmacy Building - Barts Health NHS Trust, London
  - Hammersmith Hospital, Imperial College School Of Medicine - Imperial College Healthcare NHS Trust, London
  - Royal Cornwall Hospital (RCH), Truro

IPD SHARING:
Plan to Share IPD: No